CLINICAL TRIAL: NCT07387224
Title: Study to Identify Patients With Advanced Chronic Conditions in Need of Palliative Care: Validation of the NECPAL Instrument.
Brief Title: Identification of Patients With Advanced Chronic Diseases in Need of Palliative Care
Acronym: NECPAL_HUIL
Status: Active, not recruiting | Type: Observational
Sponsor: Infanta Leonor University Hospital (Other)
Collaborators: Fundación para la Investigación e Innovación Biomédica (FIIB) del Hospital Universitario Infanta Leonor y Hospital Universitario del Sureste (Unknown)
Responsible Party: Principal Investigator, Anabel Franco Moreno, Principal Investigator, Infanta Leonor University Hospital
Other Study IDs: NECPAL_HU-Infanta Leonor
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Advanced Chronic Disease; Palliative Care; Chronic Disease; Multimorbidity; Mortality Prediction
Keywords: NECPAL tool; Palliative Care Needs; Advanced Chronic Conditions; Early Identification; Screening Tool; Observational Study; Prediction
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 38 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Cohort: Adult patients with advanced oncological and non-oncological chronic diseases hospitalized for an acute medical condition or attending a day hospital, assessed using the NECPAL screening tool as part of routine clinical care. No experimental intervention is assigned.

SUMMARY:
Patients with advanced chronic diseases often have complex health needs and may benefit from palliative care. However, many of these patients are not identified early enough to receive appropriate palliative care interventions.

This prospective observational study aims to identify hospitalized patients and patients attending a day hospital with advanced chronic conditions who have palliative care needs, using the NECPAL tool. NECPAL is a validated screening instrument designed to identify patients with advanced chronic diseases who may benefit from palliative care, based on clinical indicators, disease progression, functional decline, and health care utilization.

Adult patients with advanced oncological and non-oncological chronic diseases will be consecutively evaluated. The NECPAL tool will be applied by trained investigators as part of routine clinical assessment. Patients will be classified as NECPAL positive or NECPAL negative according to predefined criteria.

The study will estimate the proportion of patients identified as NECPAL positive, describe their clinical characteristics, and analyze whether they are receiving palliative care. Secondary objectives include comparing clinical variables, comorbidity indices, and mortality between NECPAL-positive and NECPAL-negative patients over follow-up.

The results of this study will provide information on the prevalence of palliative care needs among patients with advanced chronic diseases and support early identification strategies in hospital settings.

DETAILED DESCRIPTION:
This is a prospective, observational, analytical study designed to identify patients with advanced chronic conditions who have palliative care needs, using the NECPAL screening tool.

The study will be conducted in hospitalized patients admitted for an acute medical condition and in patients attending a day hospital. Adult patients with at least one advanced chronic oncological or non-oncological disease will be consecutively assessed during routine clinical care.

The NECPAL tool will be applied by trained investigators following the standardized methodology recommended by its developers. The assessment begins with the Surprise Question ("Would you be surprised if this patient died within the next 12 months?"). If the answer is negative, additional clinical indicators related to disease severity, functional decline, comorbidity, symptom burden, and health care utilization are evaluated. Patients will be classified as NECPAL positive or NECPAL negative according to predefined criteria.

For patients identified as NECPAL positive, information regarding current palliative care involvement will be recorded. Clinical, functional, social, and health care utilization variables will be collected from the electronic medical record as part of routine clinical documentation.

Secondary analyses will compare NECPAL-positive and NECPAL-negative patients in terms of comorbidity, functional status, and mortality. Mortality will be assessed during follow-up using hospital records and, when necessary, telephone contact.

The study aims to describe the prevalence of palliative care needs in patients with advanced chronic diseases, evaluate the alignment between identified needs and current palliative care provision, and support early identification of patients who may benefit from palliative care in hospital settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Hospitalized patients admitted for an acute medical condition or patients attending a day hospital.
* Presence of at least one advanced chronic oncological or non-oncological disease.
* Ability to provide informed consent or availability of a legally authorized representative to provide consent.

Exclusion Criteria:

* Patients in the last days of life at the time of assessment.
* Patients who die during the acute hospitalization process.
* Patients with end-stage organ failure who are listed for organ transplantation.
* Patients with severe psychiatric disease that interferes with study participation.
* Patients previously included in the study during a prior hospital admission.
* Patients for whom outpatient follow-up cannot be ensured.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients with advanced oncological and non-oncological chronic diseases who are hospitalized for an acute medical condition or evaluated in a day hospital setting. Patients are consecutively assessed as part of routine clinical care and screened for palliative care needs using the NECPAL tool.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Identified as NECPAL Positive | At baseline (at the time of inclusion)
  Proportion of adult patients with advanced oncological and non-oncological chronic diseases who are identified as NECPAL positive using the NECPAL screening tool during hospital admission or day hospital assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Infanta Leonor, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the observational nature of the study and the inclusion of sensitive clinical data collected from routine care. Data sharing would require additional ethical approvals and data-sharing agreements that are not currently planned.